CLINICAL TRIAL: NCT05801991
Title: Neurolens and Contact Lens Discomfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southern California College of Optometry at Marshall B. Ketchum University (Other)
Collaborators: Neurolens Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCCOCLNeurolens
Record Dates: First submitted 2023-03-24; First posted 2023-04-06 (Actual); Results first posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-03

CONDITIONS: Contact Lens Discomfort

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Neurolens Treatment (Experimental): Participants will receive Neurolens lenses (measured with the Neurolens device while wearing their habitual contact lenses) in their study spectacles
  Interventions: Device: Neurolens
- Placebo Lens (Placebo Comparator): Participants will receive plano (no power) lenses in their study spectacles
  Interventions: Device: Placebo spectacle lens

INTERVENTIONS:
Device: Neurolens — neurolens® is a type of spectacle lens that uses contoured prism to alleviate vergence demands and fatigue at near and, therefore, encourages comfortable vision.8 This spectacle design uses the neurolens® Measurement Device (nMD) to measure eye alignment and determine the spectacle lenses that are uniquely designed for each wearer.
  Arms: Neurolens Treatment
Device: Placebo spectacle lens — Plano (no power) spectacle lenses will be assigned to the placebo group
  Arms: Placebo Lens

SUMMARY:
The objective of this study is to determine how neurolens® influences contact lens discomfort in uncomfortable myopic soft contact lenses wearers. It is hypothesized that uncomfortable soft contact lens wearers are experiencing some level of discomfort associated with increased vergence demand when looking at near targets and will experience discomfort relief when wearing neurolens® over their habitual soft contact lenses. Uncomfortable, myopic soft contact lens wearers will be recruited. Each participant will be masked and randomly assigned a placebo pair of spectacles or a neurolens® spectacle pair for approximately one month. A prospective, randomized clinical trial will be performed. Participants and investigators will be masked to the treatment.

DETAILED DESCRIPTION:
Discomfort is the primary reason for contact lens dissatisfaction and discontinuation. Symptoms of contact lens discomfort are often attributed to dryness; however, severity of dry eye and discomfort symptoms is not correlated with clinical dry eye severity. When clinical signs of contact lens discomfort and dryness misalign with symptom severity, the possibility of an under-recognized etiology must be considered.

Symptoms associated with contact lens discomfort are similar to symptoms reported with binocular vision disorders and accommodative and vergence strain. Eyestrain, fatigue, and increased/more frequent end-of-day symptoms are noted by patients in both groups of conditions. It has been reported that uncomfortable contact lens wearers have an unusually high prevalence of binocular vision disorders and clinical signs. Basic optical calculations show that myopes must converge and accommodate more when corrected with contact lenses versus spectacles, so it is reasonable to hypothesize that a myopic contact lens wearer may experience eyestrain and discomfort associated with vergence fatigue while wearing contact lenses, but not while wearing single vision spectacles.

neurolens® is a type of spectacle lens that uses contoured prism to alleviate vergence demands and fatigue at near and, therefore, encourages comfortable vision. This spectacle design uses the neurolens® Measurement Device (nMD) to measure eye alignment and determine the spectacle lenses that are uniquely designed for each wearer. Acknowledging that some amount of contact lens discomfort may be caused by vergence fatigue, it is possible that uncomfortable contact lens wearers who wear neurolens® over their contact lenses will achieve discomfort relief.

The objective of this study is to determine how neurolens® influences contact lens discomfort in uncomfortable myopic soft contact lenses wearers. Investigators hypothesize that uncomfortable soft contact lens wearers are experiencing some level of discomfort associated with increased vergence demand when looking at near targets and will experience discomfort relief when wearing neurolens® over their habitual soft contact lenses. Uncomfortable, myopic soft contact lens wearers will be recruited. Each participant will be masked and randomly assigned a placebo pair of spectacles or a neurolens® spectacle pair for approximately one month. A prospective, randomized clinical trial will be performed. Participants and investigators will be masked to the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Uncomfortable soft contact lens wearers (CLDEQ-8 ≥ 17 points)
* Adult, pre-presbyopic age range (18 - 35 years)
* Visual acuity of 20/25 or better in each eye with habitual contact lenses
* Soft, spherical or low toric, single vision soft contact lens wearer:

  * Habitual contact lens sphere power -0.75 D or more myopic
  * Habitual contact lens are spherical design or have 1.75 D or less of cylinder correction
  * Habitual soft contact lenses are single vision design
  * Valid contact lens prescription at the date of the baseline
  * No significant subjective over-refraction in either eye with habitual soft contact lenses
* No significant subjective over-refraction in either eye with habitual soft contact lenses

  * Sphere: ≤ 0.50 D myopia, ≤ 0.50 D hyperopia
  * Cylinder: ≤ 0.75 D
* Valid measurement on the neurolens® Measurement Device (nMD2)

  * A numerical neurolens value
  * No low Measurement Quality Index (MQI) < 0.8 or convergence excess

Exclusion Criteria:

* History of ocular surgery
* History of ocular disease, amblyopia, strabismus, or vision therapy
* History of neurolens or prism spectacle correction
* History of significant vertical phoria or vertical phoria correction
* Current ocular medication use
* Significant signs of dry eye:

  * > Grad 1 ocular surface staining
  * Schirmer scores < 7 mm
  * Tear break up time < 7 seconds
* Signs of inappropriate fit or surface of soft contact lenses

  * Insufficient movement centration, and/or coverage
  * Significant lens deposits
  * Signs of corneal or conjunctival contact-lens related complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Rueff, OD, PhD, Principal Investigator — Marshall B. Ketchum University
Locations (1):
- The Southern California College of Optometry at Marshall B. Ketchum University, Fullerton, California, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers at this time.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Neurolens Treatment | Placebo Lens
Started | 15 | 15
Completed | 14 | 15
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neurolens Treatment | Placebo Lens | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.57 (2.14) | 26.20 (3.26) | 25.41 (2.85)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Male | 10 | 13 | 23
  Gender: Female | 2 | 2 | 4
  Gender: Chose not to declare | 2 | 0 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 14 | 15 | 29
Mean Contact Lens Wear Time (hours/day) [Mean (Standard Deviation); unit: hours/day] | 10.79 (3.58) | 10.80 (3.63) | 10.79 (3.48)
Mean Contact Lens Wear Time (days/week) [Mean (Standard Deviation); unit: days/week] | 5.79 (1.25) | 5.53 (1.46) | 5.66 (1.32)

OUTCOME MEASURES:

1. Primary Outcome: Change in Contact Lens Discomfort
Description: Change in contact lens discomfort measured by the Contact Lens Dry Eye Questionnaire-8 (CLDEQ-8), Score range: 0 - 37 points, Higher scores indicate worse symptoms
Time Frame: Baseline and 30-35 days
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Neurolens Treatment | Placebo Lens
Number analyzed (Participants) | 14 | 15
Scores on a scale | -4.94 (3.84) | -8.67 (5.03)

2. Secondary Outcome: Change in Convergence Insufficiency Symptoms
Description: Change in convergence insufficiency symptoms measured by the Convergence Insufficiency Symptom Survey (CISS), Score range 0 - 60 points, Higher scores indicate worse symptoms
Time Frame: Baseline and 30-35 days
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Neurolens Treatment | Placebo Lens
Number analyzed (Participants) | 14 | 15
Scores on a scale | -8.86 (7.63) | -8.93 (9.58)

3. Secondary Outcome: Change in Headache Symptoms
Description: Change in headache symptoms measured by the Headache Impact Test (HIT-6), Score range: 36 - 78 points, Higher scores indicate worse symptoms
Time Frame: Baseline and 30-35 days
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Neurolens Treatment | Placebo Lens
Number analyzed (Participants) | 14 | 15
Scores on a scale | -3.14 (9.69) | -9.73 (9.63)

4. Secondary Outcome: Change in Dry Eye Symptoms
Description: Change in dry eye symptoms measured by the Standard Patient Evaluation of Eye Dryness (SPEED) survey, Score range: 0 - 28 points, Higher scores indicated worse symptoms
Time Frame: Baseline and 30-35 days
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Neurolens Treatment | Placebo Lens
Number analyzed (Participants) | 14 | 15
Scores on a scale | -4.29 (4.30) | -6.67 (4.47)

ADVERSE EVENTS:
Time Frame: Baseline and 30-35 days
Arm/Group | Neurolens Treatment | Placebo Lens
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-10): https://cdn.clinicaltrials.gov/large-docs/91/NCT05801991/Prot_SAP_000.pdf